CLINICAL TRIAL: NCT03778697
Title: Safety and Efficacy of Endoscopic Sleeve Gastroplasty in Obese Children and Adolescents
Brief Title: Endosleeve in Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: New You Medical Center (Unknown)
Responsible Party: Principal Investigator, Aayed Alqahtani, Professor of Surgery, Director of Obesity Chair, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KingSaudU2018
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent Endosleeve (Experimental): Patients who will undergo endoscopic sleeve gastroplasty
  Interventions: Procedure: Endoscopic Sleeve Gastroplasty

INTERVENTIONS:
Procedure: Endoscopic Sleeve Gastroplasty — Endoscopic full-thickness suture system to plicate the greater curvature of the stomach
  Other Names: Endosleeve

SUMMARY:
In this study, the investigators assess the safety and efficacy of endoscopic sleeve gastroplasty in adolescents with obesity.

DETAILED DESCRIPTION:
Endoscopic bariatric therapy (EBT) is an emerging, rapidly evolving field that aims to serve as a middle ground between safe, albeit poorly effective medical weight loss strategies and drastic but effective bariatric surgery. Endoscopic sleeve gastroplasty (ESG) is a procedure that restricts the stomach to a sleeve-like configuration by utilizing full-thickness sutures that plicate the greater curvature of the stomach. Emerging data from adult populations shows an acceptable safety, tolerability and efficacy profile. Based on analysis that confirmed the safety and efficacy of ESG in adult patients who undergo the procedure under a standardized protocol and clinical care pathway, the investigators planned to study its effects on adolescents in a specialized center that offers surgical, endoscopic, and medical management of obesity under a standardized protocol and care pathway.

ELIGIBILITY:
Inclusion Criteria:

* BMI that is >120% of the 95th percentile for age and gender
* Written informed assent/consent, with concomitant parental consent for patients aged ≤17 years

Exclusion Criteria:

* Age <10 years
* Age >21 years
* Presence of large hiatal hernia
* Previous gastric surgery
* Cognitive impairment

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Weight Loss | One year
  % total weight loss
Adverse events | One year
  Adverse events, including hospitalization, or unplanned intervention

CONTACTS AND LOCATIONS:
Overall Officials: Aayed R Alqahtani, MD FRCSC FACS, Principal Investigator — King Saud University
Locations (1):
- New You Medical Center, Riyadh, Central Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alqahtani A, Elahmedi M, Alqahtani YA, Al-Darwish A. Endoscopic Sleeve Gastroplasty in 109 Consecutive Children and Adolescents With Obesity: Two-Year Outcomes of a New Modality. Am J Gastroenterol. 2019 Dec;114(12):1857-1862. doi: 10.14309/ajg.0000000000000440. PMID 31658128